CLINICAL TRIAL: NCT03994328
Title: An Observational, Prospective, Multinational, Multicentre Study Comparing the Effectiveness of Safinamide, Rasagiline and Other "Standard Of Care" as Add-On Therapy to Levodopa (L-Dopa) in Parkinson's Disease (Pd) Fluctuating Patients
Brief Title: An Observational Study on Safinamide, Rasagiline and Other Standard of Care in PD
Acronym: SUCCESS
Status: Completed | Type: Observational
Sponsor: Zambon SpA (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: Z7219N04
Record Dates: First submitted 2019-06-18; First posted 2019-06-21 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's; PD; Safinamide; Rasagiline; Levodopa; L-DOPA; Fluctuating Patients; Add-on Therapy; PDQ; UPDRS; NRS; quality of life; observational
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: 500 patients already receiving safinamide (50 or 100 mg/day) as add-on to L-dopa for no more than 2 months.
- Group 2: 500 patients receiving rasagiline 1 mg/day as add-on to L-dopa for no more than 2 months.
- Group 3: 235 patients receiving other SoC drugs as add-on to L-dopa for no more than 2 months.

SUMMARY:
The purpose of this study is to evaluate how safinamide, rasagiline and other SoC drugs are associated with the quality of life of PD patients by means of the Parkinson's Disease Questionnaire (PDQ)-39 items.

DETAILED DESCRIPTION:
Safinamide is an alpha-aminoamide derivative, structurally unrelated to any other drug for the treatment of PD, with a dual mechanism of action (dopaminergic and non-dopaminergic). In particular, it is a potent, selective and reversible MAO-B inhibitor, and it is a glutamate modulator through the sodium channels blockade.

Safinamide has been approved in Europe for the treatment of mid- to late-stage patients with idiopathic PD and fluctuations as add-on therapy to a stable dose of levodopa (alone or in combination with other PD medications).

Rasagiline is an irreversible MAO-B inhibitor, with unknown activity on other neurotransmitters. Rasagiline has been approved in Europe for the treatment of idiopathic PD as monotherapy or as add-on to levodopa in patients with end of dose fluctuations.

The aim of this observational study is to evaluate the effectiveness of safinamide, rasagiline and other "standard of care" (SoC) drugs when prescribed in clinical routine as add-on to L-dopa in terms of quality of life, improvement of chronic pain, change in Anti-Parkinson treatment (modification of doses, addition or withdrawal or other Anti-Parkinson drugs, etc.), use of concomitant pain-killer medications, compliance to the PD treatment, hospitalizations and use of other healthcare resources, and number of lost working days.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders ≥ 18 years of age, with a clinical diagnosis of idiopathic PD according to UK Brain Bank diagnostic criteria (12) for whom safinamide, rasagiline or any other anti-Parkinson drugs are prescribed according to the current Summary of Product Characteristics (SmPC).
* Willing to participate in the study and able to understand and sign the written informed consent form.
* Patients on a stable anti-Parkinson therapy, always including L-dopa + dopa-decarboxylase inhibitor (DDI), with or without other anti-Parkinson medications.
* Patients must be treated with safinamide, rasagiline or other SoC drugs as add-on to L-dopa for no more than 2 months prior to the baseline visit, according to the clinical practice.

Exclusion Criteria:

* Patients with any form of Parkinsonism other than idiopathic PD.
* Patients for whom safinamide, rasagiline or any other anti-Parkinson drug are contraindicated according to the current SmPC.
* Patients known to be pregnant.
* Patients treated with safinamide or rasagiline who receive other concomitant MAO-B inhibitors.
* Patients treated with other SoC drugs who receive safinamide or rasagiline.
* Previous participation in a clinical trial with an investigational drug or medical device in the 3 months prior to the baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 1235 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The change from baseline to the end of study of the PDQ-39 total score. | The validated PDQ-39 assesses health-related quality improvement (Qi); an improvement in Qi corresponds to a decrease of the PDQ-39 total score.
  Over a period of 12 months

SECONDARY OUTCOMES:
PDQ-39 total score | 6 months
  The change from baseline to 6 months in the PDQ-39 total score.
PDQ-39 sub-scores (domains and single items) | 6 and 12 months
  The change from baseline to 6 months and to the end of study (12 months) in the PDQ-39 sub-scores (domains and single items)
UPDRS III score | 6 and 12 months
  The change from baseline to 6 months and to the end of study (12 months) in the UPDRS III score.
NRS. | 6 and 12 months
  The change from baseline to 6 months and to the end of study (12 months) in the NRS
anti-Parkinson drugs number | 6 and 12 months
  The change in anti-Parkinson drugs number from baseline to 6 months and to the end of the study (12 months).
new anti-Parkinson drugs | 6 and 12 months
  The introduction of new anti-Parkinson drugs, withdrawal, augmentation and decrease at 6 and 12 months, respectively.
The use of concomitant pain-killer medications | 6 and 12 months
  The use of concomitant pain-killer medications at 6 and 12 months, respectively.
number of pain-killer medications | 6 and 12 months
  The change in the number of pain-killer medications from baseline to 6 months and to the end of the study (12 months).
new pain-killer medications and daily dosage of pain-killer medications | 6 and 12 months
  The introduction of new pain-killer medications, withdrawal, augmentation, decrease and daily dosage of pain-killer medications at 6 and 12 months, respectively.
Healthcare resources | 6 and 12 months
  The use of healthcare resources from baseline to 6 months and to the end of study (12 months): number of and reason for hospitalizations, number of hospitalization days, number of visits to the emergency room, number of visits to PD specialists, number of diagnostic exams, number of rehabilitation visits.
number of working-days lost | 6 and 12 months
  The number of working-days lost from baseline to 6 months and to the end of study (12 months).
Safety Endpoints | 6 and 12 months
  The nature, frequency, severity, relationship (to study drug), actions taken, and outcome of adverse events (AEs) and serious adverse events (SAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Cattaneo, Study Director — Zambon Group
Locations (3):
- Praxis Dr. med. Kirsten Hahn, Berlin, Germany
- Università degli Studi G. D'Annunzio, Chieti, Italy
- Corporacio Sanitaria Parc Tauli, Sabadell, Spain

REFERENCES:
- [Background] Poewe W, Seppi K, Tanner CM, Halliday GM, Brundin P, Volkmann J, Schrag AE, Lang AE. Parkinson disease. Nat Rev Dis Primers. 2017 Mar 23;3:17013. doi: 10.1038/nrdp.2017.13. PMID 28332488
- [Background] Fox SH. Non-dopaminergic treatments for motor control in Parkinson's disease. Drugs. 2013 Sep;73(13):1405-15. doi: 10.1007/s40265-013-0105-4. PMID 23917951
- [Background] Wirdefeldt K, Adami HO, Cole P, Trichopoulos D, Mandel J. Epidemiology and etiology of Parkinson's disease: a review of the evidence. Eur J Epidemiol. 2011 Jun;26 Suppl 1:S1-58. doi: 10.1007/s10654-011-9581-6. Epub 2011 May 28. PMID 21626386
- [Background] Connolly BS, Lang AE. Pharmacological treatment of Parkinson disease: a review. JAMA. 2014 Apr 23-30;311(16):1670-83. doi: 10.1001/jama.2014.3654. PMID 24756517
- [Background] Fabbrini G, Brotchie JM, Grandas F, Nomoto M, Goetz CG. Levodopa-induced dyskinesias. Mov Disord. 2007 Jul 30;22(10):1379-1389. doi: 10.1002/mds.21475. PMID 17427940
- [Background] Chaudhuri KR, Schapira AH. Non-motor symptoms of Parkinson's disease: dopaminergic pathophysiology and treatment. Lancet Neurol. 2009 May;8(5):464-74. doi: 10.1016/S1474-4422(09)70068-7. PMID 19375664
- [Background] Neff C, Wang MC, Martel H. Using the PDQ-39 in routine care for Parkinson's disease. Parkinsonism Relat Disord. 2018 Aug;53:105-107. doi: 10.1016/j.parkreldis.2018.05.019. Epub 2018 May 17. PMID 29853294
- [Background] Caccia C, Maj R, Calabresi M, Maestroni S, Faravelli L, Curatolo L, Salvati P, Fariello RG. Safinamide: from molecular targets to a new anti-Parkinson drug. Neurology. 2006 Oct 10;67(7 Suppl 2):S18-23. doi: 10.1212/wnl.67.7_suppl_2.s18. PMID 17030736
- [Background] ISPE. Guidelines for good pharmacoepidemiology practices (GPP). Pharmacoepidemiol Drug Saf. 2008 Feb;17(2):200-8. doi: 10.1002/pds.1471. No abstract available. PMID 17868186
- [Background] Hoehn MM, Yahr MD. Parkinsonism: onset, progression and mortality. Neurology. 1967 May;17(5):427-42. doi: 10.1212/wnl.17.5.427. No abstract available. PMID 6067254
- [Background] Peto V, Jenkinson C, Fitzpatrick R, Greenhall R. The development and validation of a short measure of functioning and well being for individuals with Parkinson's disease. Qual Life Res. 1995 Jun;4(3):241-8. doi: 10.1007/BF02260863. PMID 7613534
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] Morisky DE, Ang A, Krousel-Wood M, Ward HJ. Predictive validity of a medication adherence measure in an outpatient setting. J Clin Hypertens (Greenwich). 2008 May;10(5):348-54. doi: 10.1111/j.1751-7176.2008.07572.x. PMID 18453793
- [Derived] Lawn T, Rukavina K, Malcangio M, Howard M, Chaudhuri KR. Response to Mylius et al. Pain. 2022 Mar 1;163(3):e496-e497. doi: 10.1097/j.pain.0000000000002445. No abstract available. PMID 35148289